CLINICAL TRIAL: NCT04135755
Title: The Spine Kinematics and Center of Pressure Excursion During Functional Task in Scoliosis and Vertebral Compression Fractures Subjects
Brief Title: The Spine Kinematics and Center of Pressure Excursion During Functional Task Vertebral Compression Fractures Subjects
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Hungkuang University (Other)
Responsible Party: Sponsor
Other Study IDs: CF15027A
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2015-02

CONDITIONS: Posture; Vertebral Compression Fracture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- vertebral compression fracture: No drugs intervention
  Interventions: Other: no drug intervention
- older adult without spinal deformity: No drugs intervention
  Interventions: Other: no drug intervention
- young adults: No drugs intervention
  Interventions: Other: no drug intervention

INTERVENTIONS:
Other: no drug intervention — no drug or treatment intervention

SUMMARY:
This study aimed to assess the sensory and kinematic components of the limits of stability (LOS) test in patients with vertebral compression fracture (VCF) .

DETAILED DESCRIPTION:
This study enrolled adults with VCF (VCF group), older adult without spinal deformity (NE group), and young adults (NY group). The Biodex balance system was employed to calculate the balance score and the LOS of participants. An inertia motion system was used to record kinematic data. The center of pressure (COP) signals of postural stability and LOS were used to calculate the frequency power spectrum for interpreting the sensory component.

ELIGIBILITY:
Vertebral compression fracture Inclusion Criteria:

older than 65 years osteoporosis diagnosed by a bone mineral density test of the lumbar spine (T-score < -2.5; T: peak bone mass) thoracic-lumbar VCF on radiography without displacement

Vertebral compression fracture Exclusion Criteria:

other spinal diseases that might also cause back pain (such as scoliosis, lumbar spondylolisthesis, lumbar disk disease, and spinal stenosis) a history of diabetes a history of neurological disease (such as cerebral vascular disease, peripheral neuropathy and vestibular disease).

Control Inclusion Criteria:

None the control participants had evidence of gait, postural, or spine disorders.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolled 13 adults with VCF, 13 older adult without spinal deformity, and 13 young adults.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2016-08-22 (Actual)

PRIMARY OUTCOMES:
Postural Stability | 90 second
  A balance system was employed to calculate the standing posture sway score.A high score was indicative of excessive movement during the test and thus, poor stability. The range of value was 0.3- 4.1.
limits of stability | 1-2 minutes
  patients shift their center of gravity from the center target to a blinking target and back to the center target.This process was repeated for each of the 9 targets. A high score was indicative of fine direction control.The range of value was 21- 66.
Kinematic Data | 5 minutes
  The movements of the head, upper spine, lower spine, pelvis,hip, thigh, and knee were measured using 6 inertial measurement units.
timed up-and-go test | 90 second
  sit-stand-walk-180° turning-walk and sitting down task

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Tsu Chang, phD, Principal Investigator — Taichung Veterans General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lynn SG, Sinaki M, Westerlind KC. Balance characteristics of persons with osteoporosis. Arch Phys Med Rehabil. 1997 Mar;78(3):273-7. doi: 10.1016/s0003-9993(97)90033-2. PMID 9084349
- [Derived] Kuo FC, Chang ST, Liao YY, Lee CH. Center of Pressure Trace and Sensory Components of the Limits of Stability Test in Older Adults With Vertebral Compression Fractures. J Geriatr Phys Ther. 2020 Jan/Mar;43(1):24-31. doi: 10.1519/JPT.0000000000000201. PMID 29923897